CLINICAL TRIAL: NCT05783011
Title: The Effects of Electroacupuncture on Postoperative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Didem OZKAL EMINOGLU (Other)
Responsible Party: Sponsor-Investigator, Didem OZKAL EMINOGLU, assistant professor, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2022
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Periodontal Diseases; Periodontitis; Acupuncture; Electroacupuncture
Keywords: Periodontitis; Acupuncture; Electroacupuncture
MeSH Terms: conditions — Periodontal Diseases; Periodontitis | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EA (electroacupuncture) (Experimental): Individuals who underwent electroacupuncture before and after flap surgery
  Interventions: Procedure: Electroacupuncture; Procedure: periodontal flap surgery
- Control (Active Comparator): Individuals who have undergone flap surgery only
  Interventions: Procedure: periodontal flap surgery

INTERVENTIONS:
Procedure: Electroacupuncture — Electroacupuncture was applied bilaterally to the LI4, ST5 and ST6 acupuncture points before and after periodontal flap surgery
  Arms: EA (electroacupuncture)
Procedure: periodontal flap surgery — periodontal flap surgery

SUMMARY:
In this study,the investigators aimed to examine the effect of electroacupuncture application on the amount of pain felt by patients after periodontal surgery.

The main question it aims to answer is there any efficiacy of electroacupuncture application on postoperative pain reduction.

Participants will get periodontal flap surgery treatment with/without electroacupuncture

Researchers will compare EA and control groups to see if there is any relationship between acupuncture application and postoperative pain

DETAILED DESCRIPTION:
Postoperative pain is an acute pain that begins with surgical trauma and decreases over time with tissue healing. The level of pain and discomfort felt varies from person to person. The patient's sex and age, physiological and psychological structure, operation area, duration of surgery, premedication, type of anesthetic used, postoperative complications and several other environmental factors can affect this level. After the operation, especially within 48 hours, the pain increases and gradually decreases. Postoperative pain may cause an increase in anxiety and general fear and concern. The stress level caused by surgical trauma in the patient delays recovery and increases mortality and morbidity.

Electroacupuncture (EA) applies electrical stimulation current to needles placed on acupuncture points. It is mainly used to relieve pain and provide operative analgesia.

No study has been found in the literature on the pain-reducing functionality of acupuncture applications in periodontal surgical treatments. In this study, the investigators aimed to examine the effect of electroacupuncture application on the amount of pain felt by patients after periodontal surgery.

ELIGIBILITY:
Inclusion Criteria:

* absence of any systemic disease,
* pregnancy or breast feeding;
* not receiving anti-inflammatory drug therapy in the last 6 months, chemotherapy or radiotherapy;
* having 6 mm or more probable pocket depth and clinical attachment loss in at least 4 or more teeth when called for control 6 weeks after Phase I treatment

Exclusion Criteria:

* Having a systemic disease such as cardiovascular, diabetes, hypertension, thyroid organ pathologies, chronic kidney failure
* pregnant/breastfeeding
* medication for any reason
* smoker/tobacco user
* other periodontal disease other than periodontitis
* chronic inflammatory disease (COPD, asthma)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 7 days
  The Visual Analogue Scale consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be')

SECONDARY OUTCOMES:
Postoperative analgesic requirement | 7 days
  the number of analgesic requirements taken by patients after periodontal surgery.

CONTACTS AND LOCATIONS:
Overall Officials: DİDEM ÖZKAL EMİNOĞLU, Study Director — Ataturk University
Locations (1):
- Atatürk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided